CLINICAL TRIAL: NCT01282060
Title: Association Between Glycaemic Control and Morbi/Mortality After 5 Years of Follow-up in Type 2 Diabetic Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Association Pour la Recherche en Diabetologie et en Geriatrie (Other)
Collaborators: Novo Nordisk A/S (Industry); Umanis (Industry)
Responsible Party: Sponsor
Other Study IDs: CRO0662-1
Record Dates: First submitted 2011-01-21; First posted 2011-01-24 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2017-01

CONDITIONS: Type 2 Diabetes
Keywords: HBA1C; DIABETES-RELATED COMPLICATIONS; GLYCAEMIC BALANCE
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to asses the link between glycaemic balance (summarised by HBA1C LEVEL) and specific causes of death.

DETAILED DESCRIPTION:
The GERODIAB study is the first prospective, longitudinal follow-up cohort study, the main aim of which is to assess the link between glycaemic balance (evaluated on the basis of HbA1c levels) and total mortality at 5 years in diabetic patients aged 70 and over, and suffering from type 2 diabetes. An extension to 10 years is considered given the innovative features of this cohort follow-up procedure.

The secondary endpoints are as follows:

* To assess the link between glycaemic balance and the mortality rate with specific causes.
* To assess the link between glycaemic balance and the onset of or change in diabetes-related complications: cardiovascular diseases, change in renal function, diabetic retinopathy, peripheral neuropathy, perforating ulcer of the foot and acute metabolic complications.
* To assess the link between glycaemic balance and nutritional status, the onset of or changes in cognitive disorders and a loss of autonomy.
* To specify the role of other cardiovascular risk factors combined with glycaemic balance, in mortality, diabetes-related complications, cognitive disorders and loss of autonomy.

ELIGIBILITY:
Inclusion Criteria:

* Patient with type 2 diabetes, aged 70 and over,
* Patient having received medicinal or non-medicinal treatment (in the case of diabetics treated with insulin, the length of time between diagnosis of diabetes and the onset of insulin therapy will be at least 2 years),
* Diabetes diagnosed for at least one year,
* Patient with autonomy defined by a score greater than or equal to 3/6 on the ADL scale,
* Patient who can be monitored during hospital or private consultations over the next 10 years,
* Patient who did not refuse to take part in the study after receiving information on the study (Patient Information Leaflet), Patients are monitored in the hospital or private sector throughout France.

Exclusion Criteria:

* Patient with type 1 diabetes,
* Patient with secondary diabetes (mainly corticosteroid-induced),
* Patient with a loss of autonomy defined by a score of less than 3/6 on the ADL scale,
* Patient who cannot be monitored in the months or years to come,
* Patient in an acute situation (transient exclusion criterion),
* Patient expressing their refusal to participate in the study.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: * Patients suffering from type 2 diabetes and aged 70 and over.
  * Having received medicinal or non-medicinal therapy (in the case of diabetics treated with insulin, the lengh of time between diagnosis of diabtees and the introduction of insulin therapy is at least 6 months).
  * Suffering from type 2 diabetes at least one year.
  * With autonomy defined by a score greater than or equal to 3/6 on the ADL scale and able of being followed-up during hospital or private consultations over the next 5 years.
  * Patients who did not refuse to participate in the study after receiving information on the study (Patient Information Leaflet).
  The patient are monitored in the hospital or private sector throughout Metropolitan France.
Sampling Method: Probability Sample
Enrollment: 986 (Actual)
Dates: Start 2009-03; Primary Completion 2016-04 (Actual); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Link between HbA1c level and the overall mortality rate at 5 years. | 5 years
  The primary endpoint is to assess the link between glycaemic balance (assessed on the basis of the HbA1c level) and the overall mortality rate at 5 years for patients of 70 and over suffering from type 2 diabetes.

SECONDARY OUTCOMES:
Link between HbA1c level and specific causes of death. | 5 years
  To assess the link between glycaemic balance (summarised by HbA1c level) and specific causes of death.
Link between HbA1c level and the onset of or changes in diabetes-related complications | 5 years
  To assess the link between glycaemic balance (summarised by HbA1c) and the onset of or changes in diabetes-related complications: - cardiovascular diseases (coronary failure, heart failure, cerebrovascular accidents, arteriopathy obliterans of the lower limbs), - change in renal function, diabetic retinopathy, peripheral neuropathy, perforating ulcer of the foot, acute metabolic complications (hypoglycaemia, diabetic ketoacidosis, hyperosmolarity).
Link between HbA1c level and nutritional status. | 5 years
  To assess the link between glycaemic balance and nutritional status.
Link between HbA1c level and the onset of or changes in cognitive disorders. | 5 years
  To assess the link between glycaemic balance and the onset of or changes in cognitive disorders.
Link between HbA1c level and loss of autonomy. | 5 years
  To assess the link between glycaemic balance and loss of autonomy.
Role of other cardiovascular risk factors | 5 years
  To specify the role of other cardiovascular risk factors (primarily, arterial hypertension, dyslipidaemia and obesity) in association with glycaemic balance on the mortality rate, diabetes-related complications, cognitive disorders and loss of autonomy.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Doucet J, Verny C, Bordier L, Rekik A, Zulfiqar AA, Bezerra CB, Bauduceau B. Evolution in geriatric syndromes and association with survival over 5 years in the GERODIAB cohort of older French diabetic patients. Eur Geriatr Med. 2021 Jun;12(3):619-625. doi: 10.1007/s41999-020-00425-9. Epub 2020 Nov 22. PMID 33225383
- [Derived] Doucet J, Verny C, Balkau B, Scheen AJ, Bauduceau B. Haemoglobin A1c and 5-year all-cause mortality in French type 2 diabetic patients aged 70 years and older: The GERODIAB observational cohort. Diabetes Metab. 2018 Dec;44(6):465-472. doi: 10.1016/j.diabet.2018.05.003. Epub 2018 May 18. PMID 29859993
- [Derived] Bauduceau B, Le Floch JP, Halimi S, Verny C, Doucet J; SFD/SFGG Intergroup. Cardiovascular Complications Over 5 Years and Their Association With Survival in the GERODIAB Cohort of Elderly French Patients With Type 2 Diabetes. Diabetes Care. 2018 Jan;41(1):156-162. doi: 10.2337/dc17-1437. Epub 2017 Nov 7. PMID 29113984